CLINICAL TRIAL: NCT00285103
Title: An Open-labelled, International, Multicenter, Dose Escalating, Phase I/II Study of SPC2996,an LNA Antisense Molecule Against Bcl-2, in Patients With Relapsed or Refractory Chronic Lymphocytic Leukaemia
Brief Title: SPC2996 in Chronic Lymphocytic Leukaemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Santaris Pharma A/S (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPC2996-101
Record Dates: First submitted 2005-09-12; First posted 2006-02-01 (Estimated); Last update posted 2011-02-02 (Estimated); Status verified 2011-02

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Antisense, mRNA antagonist, Bcl-2, CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: SPC2996

SUMMARY:
The purpose of this study is to determine whether SPC2996 is effective and safe in the treatment of Chronic Lymphocytic Leukaemia (CLL)

DETAILED DESCRIPTION:
Chronic Lymphocytic Leukaemia (CLL) is the most common leukaemia in adults in the US and most of Western Europe. Many patients suffering from CLL have tumour cells expressing high amounts of Bcl-2 protein. Since over expression of Bcl-2 inhibits apoptosis, it is possible that this gene participates in the pathogenesis of CLL. By lowering the Bcl-2 protein in these tumour cells the cells may go into apoptosis due to changed balance in pro- and anti apoptotic proteins and thereby it might be possible to induce a tumour response.

The study is an open-labelled, international, multicenter, dose escalating phase I/II study where patients receive 6, 3, 2 or 1 dose(s) of SPC2996, a LNA antisense molecule against Bcl-2, over a period of up to 2 weeks, and are followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* patients with relapsed or refractory Chronic Lymphocytic Leukaemia requiring therapy
* screening blood sample must show circulating lymphocyte count of more then 5 x 109/L and circulating lymphocytes expressing the phenotype CD5+CD20+CD23+.
* The PCR Bcl-2 m-RNA level must be positive
* the patients must be 18 years or older and have given informed consent.

Exclusion Criteria:

* previous treatment with rituximab, alemtuzumab or autologous stem cell transplantation within 6 months prior to Visit 1 or allogeneic stem cell transplantation at any time
* patients that received anti-cancer therapy, glucocorticoids or radiotherapy within 4 weeks prior to Visit 1 and patients with known or suspected transformation of CLL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2005-06; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Change in Bcl-2 m-RNA levels | from Day 0 to Day 13

SECONDARY OUTCOMES:
Change in Bcl-2 protein expression. Change in Bcl-2 m-RNA levels (and other parameters) | from Day 0 to Day 14 and during study respectively

CONTACTS AND LOCATIONS:
Overall Officials: Betrand Coiffier, Prof. MD, Principal Investigator — Centre Hospitalier Lyon Sud, Lyon, France
Locations (12):
- Holden Comprehensive Cancer Center, Univ. of Iowa, Iowa City, Iowa, United States
- Denmark (3):
  - Rigshospitalet, Copenhagen
  - KAS Herlev, Herlev
  - Vejle Sygehus, Vejle
- France (4):
  - Service d'HématologieCentre Hospitalier Lyon-Syd, Lyon, Cedex
  - Bruno Cazin, Lille
  - Mauricette Michellet, Lyon
  - Centre Henri Becquerel, Rouen
- United Kingdom (4):
  - Leeds General Infirmary, Leeds
  - MRC Toxicology Unit, University of Leicester, Leicester
  - Christie Hospital NHS Trust, Manchester
  - The Royal Marsden NHS Foundation Trust, Surrey